CLINICAL TRIAL: NCT05812014
Title: A Multi-center, Randomized, Blinded, Placebo-controlled, Phase 3 Clinical Study to Evaluate the Efficacy, Safety and Immunogenicity of SARS-CoV-2 Bivalent mRNA Vaccine (LVRNA021) as Booster in Participants Aged 18 Years and Older Who Completed Primary/1 Booster Dose(s) of SARS-CoV-2 Vaccination
Brief Title: Clinical Trail of SARS-CoV-2 Bivalent mRNA Vaccine (LVRNA021) in Participants Aged 18 Years and Older
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AIM Vaccine Co., Ltd. (Industry)
Collaborators: LiveRNA Therapeutics Inc. (Unknown); Ningbo Rongan Biological Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LVRNA021-III-01
Record Dates: First submitted 2023-04-10; First posted 2023-04-13 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-01

CONDITIONS: SARS-CoV-2
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Vaccine Group (Experimental)
  Interventions: Biological: SARS-CoV-2 Bivalent mRNA vaccine (LVRNA021)
- Control Group (Placebo Comparator)
  Interventions: Drug: 0.9% sodium chloride solution

INTERVENTIONS:
Biological: SARS-CoV-2 Bivalent mRNA vaccine (LVRNA021) — One dose was administered by intramuscular injection, 100μg，1.0ml/dose
  Arms: Study Vaccine Group
Drug: 0.9% sodium chloride solution — One dose was administered by intramuscular injection, 1.0ml/dose
  Arms: Control Group

SUMMARY:
This is a multi-center, randomized, blinded, placebo-controlled, phase 3 clinical study to evaluate the efficacy, safety and immunogenicity of SARS-CoV-2 bivalent mRNA vaccine (LVRNA021) as booster in participants aged 18 years and older who completed primary/1 booster dose(s) of SARS-CoV-2 vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and older;
2. Understand the content of the ICF, and voluntarily sign the ICF (If the participant is unable to sign the ICF on his/her own due to illiteracy, an impartial witness is needed);
3. Participants who are willing and able to comply with all scheduled visits, vaccination plan, laboratory tests, lifestyle considerations, and other study procedures;
4. Female participants of childbearing potential or partners of male participants: voluntarily agree to use effective contraception with their partners prior to the first vaccination and must agree to continue such precautions during the study until 3 months after booster vaccination [Effective contraception includes oral contraceptives, injectable or implantable contraception, extended-release topical contraceptives, hormonal patches, intrauterine devices (IUDs), sterilization, abstinence, condoms (for male), diaphragms, cervical caps, etc.);
5. For female participants: without childbearing potential (amenorrhea for at least 1 year or documented surgical sterilization) or have used effective contraception with a negative pregnancy test before booster vaccination in this study；
6. On the day of vaccination and 24 hours prior to vaccination, axillary temperatures<37.3°C/99.1°F;
7. Healthy participants or participants with mild underlying disease [in a stable state without exacerbation (no admission to hospital or no major adjustment to treatment regimen, etc.) for at least 3 months prior to enrollment in this study];
8. Participants who have received primary/1 booster dose(s) of SARS-CoV-2 vaccination (including primary series of inactivated vaccine, mRNA vaccine, adenovirus vaccine or 1 homologous/heterologous booster), with the last dose received at least 6 months before enrolment. Documented confirmation of prior SARS-CoV-2 vaccination receipt must be obtained prior to randomization;

Exclusion Criteria:

1. History of Severe Acute Respiratory Syndrome (SARS), Middle East Respiratory Syndrome (MERS), or other coronavirus infections at any time;
2. History of hepatitis A, hepatitis B, hepatitis C, syphilis infection based on medical inquiry.;
3. History of severe adverse reaction associated with a vaccine or drug and/or severe allergic reaction (e.g., anaphylaxis) to any component of the study intervention(s);
4. Receipt of medications intended to treat COVID-19 within 6 months;
5. Virologically confirmed SARS-CoV-2 diagnosis within 6 months before screening visit;
6. Positive nasopharyngeal/oropharyngeal swab SARS-CoV-2 RT-PCR test result at screening;
7. Positive HIV test result at screening;
8. A history or family history of convulsions, epilepsy, encephalopathy and psychosis;
9. Malignant tumors in the active phase, malignant tumors not receiving adequate treatment, malignant tumors at potential risk of recurrence during the study period;
10. Asplenia or functional asplenia, complete or partial splenectomy from any cause;
11. Individuals who receive treatment with radiotherapy or immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids (if systemic corticosteroids are administered for ≥14 days at a dose of ≥20 mg/day of prednisone or equivalent), e.g., for cancer or an autoimmune disease, or planned receipt throughout the study. Inhaled/nebulized, intra-articular, epidural, or topical (skin or eyes) corticosteroids are permitted;
12. Any other licensed vaccines given within 28 days prior to vaccination, planned administration of any other vaccines within 28 days after vaccination, or planned administration of other COVID-19 vaccines during the entire study duration;
13. Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies, from 60 days before vaccine administration, or receipt of any passive antibody therapy specific to COVID-19, from 90 days before vaccine administration, or planned receipt throughout the study;
14. Blood donation or blood loss ≥ 450 mL within 1 month prior to enrollment or planned to donate blood during the study period;
15. Participation in other studies involving study intervention within 28 days prior to study entry, and/or during the study;
16. Women who are pregnant or breastfeeding;
17. Participants deemed unsuitable for participation in this study based on the investigator's assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9800 (Estimated)
Dates: Start 2023-03-25 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Person-year incidence density of first episodes of virologically-confirmed symptomatic cases of COVID-19 | 14 days after vaccination or placebo
  The person-year incidence density of first episodes of virologically-confirmed symptomatic cases of COVID-19 of any severity meeting the case definition for the primary efficacy analysis occurring from 14 days after booster vaccination.

SECONDARY OUTCOMES:
Person-year incidence density of first episodes of virologically-confirmed moderate to severe cases of COVID-19 | 14 days after vaccination or placebo
  The person-year incidence density of first episodes of virologically-confirmed moderate to severe cases of COVID-19 from 14 days after booster vaccination meeting the case definition for the primary efficacy analysis.
Person-year incidence density of first episodes of virologically-confirmed severe cases of COVID-19 | 14 days after vaccination or placebo
  The person-year incidence density of first episodes of virologically-confirmed severe cases of COVID-19 from 14 days after booster vaccination meeting the case definition for the primary efficacy analysis.
Person-year incidence density of first episodes of virologically-confirmed cases of COVID-19 | 14 days after vaccination or placebo
  The person-year incidence density of first episodes of virologically-confirmed cases of COVID-19 leading to death from 14 days after booster vaccination meeting the case definition for the primary efficacy analysis.
Person-year incidence density of first episodes of virologically-confirmed symptomatic cases of COVID-19 for participants in different age strata (18-59 years, ≥ 60 years) | 14 days after vaccination or placebo
  The person-year incidence density of first episodes of virologically-confirmed symptomatic cases of COVID-19 of any severity occurring from 14 days after booster vaccination for participants in different age strata (18-59 years, ≥ 60 years).
Incidence of each solicited (local and systemic) AE in all participants. | within 14 days after vaccination or placebo
  Incidence of each solicited (local and systemic) AE within 14 days after booster vaccination in all participants.
Severity of each solicited (local and systemic) AE in all participants. | within 14 days after vaccination or placebo
  Severity of each solicited (local and systemic) AE within 14 days after booster vaccination in all participants.
Duration of each solicited (local and systemic) AE in all participants. | within 14 days after vaccination or placebo
  Duration of each solicited (local and systemic) AE within 14 days after booster vaccination in all participants.
Incidence of unsolicited AEs in all participants. | 0-28 days after vaccination or placebo
  Incidence of unsolicited AEs occurring 0-28 days after booster vaccination in all participants.
Severity of unsolicited AEs in all participants. | 0-28 days after vaccination or placebo
  Severity of unsolicited AEs occurring 0-28 days after booster vaccination in all participants.
Causality of unsolicited AEs in all participants. | 0-28 days after vaccination or placebo
  Causality of unsolicited AEs occurring 0-28 days after booster vaccination in all participants.
Incidence of SAEs in all participants. | within 12 months after vaccination or placebo
  Incidence of SAEs from the day of booster vaccination to 12 months after booster vaccination in all participants.
Severity of SAEs in all participants. | within 12 months after vaccination or placebo
  Severity of SAEs from the day of booster vaccination to 12 months after booster vaccination in all participants.
Incidence of AESIs in all participants. | within 12 months after vaccination or placebo
  Incidence of AESIs from the day of booster vaccination to 12 months after booster vaccination in all participants.
Severity of AESIs in all participants. | within 12 months after vaccination or placebo
  Severity of AESIs from the day of booster vaccination to 12 months after booster vaccination in all participants.
Incidence of pregnancy events in all participants. | within 12 months after vaccination or placebo
  Incidence of pregnancy events from the day of booster vaccination to 12 months after booster vaccination in all participants.
Severity of pregnancy events in all participants. | within 12 months after vaccination or placebo
  Severity of pregnancy events from the day of booster vaccination to 12 months after booster vaccination in all participants.
Causality of SAEs, AESIs, and pregnancy events in all participants. | within 12 months after vaccination or placebo
  Causality of SAEs, AESIs, and pregnancy events from the day of booster vaccination to 12 months after booster vaccination in all participants.
Geometric mean titer (GMT)of SARS-CoV-2 (Omicron subvariants) virus neutralizing antibody (live virus neutralizing assay) responses in subjects in the immunization subgroup. | 14 days,28 days,3 months and 6 months after vaccination or placebo
Seroconversion rate (SCR) of SARS-CoV-2 (Omicron subvariants) virus neutralizing antibody (live virus neutralizing assay) responses in subjects in the immunization subgroup. | 14 days,28 days,3 months and 6 months after vaccination or placebo
Geometric mean Increase (GMI) of SARS-CoV-2 (Omicron subvariants) virus neutralizing antibody (live virus neutralizing assay) responses in subjects in the immunization subgroup. | 14 days,28 days,3 months and 6 months after vaccination or placebo
GMT of S-protein IgG antibodies in subjects in the immunization subgroup. | 14 days, 28 days,3 months,6 months and 12 months after vaccination or placebo
GMI of S-protein IgG antibodies in subjects in the immunization subgroup. | 14 days, 28 days,3 months,6 months and 12 months after vaccination or placebo
SCR of S-protein IgG antibodies in subjects in the immunization subgroup. | 14 days, 28 days,3 months,6 months and 12 months after vaccination or placebo

OTHER OUTCOMES:
Person-year incidence density of first episodes of virologically-confirmed cases of COVID-19 of any severity caused by individual VOCs. | 14 days after vaccination or placebo
  The person-year incidence density of first episodes of virologically-confirmed cases of COVID-19 of any severity from 14 days after booster vaccination caused by individual VOCs.
Cellular immune subgroup:viral antigen IL-2 levels | 7 days, 14 days, 28 days and 3 months after vaccination or placebo
  Cellular immune subgroup:viral antigen IL-2 levels at 7 days, 14 days, 28 days and 3 months booster vaccination. (ELISpot assay)
Cellular immune subgroup:viral antigen IL-4 levels | 7 days, 14 days, 28 days and 3 months after vaccination or placebo
  Cellular immune subgroup:viral antigen IL-4 levels at 7 days, 14 days, 28 days and 3 months booster vaccination. (ELISpot assay)
Cellular immune subgroup:viral antigen IL-13 levels | 7 days, 14 days, 28 days and 3 months after vaccination or placebo
  Cellular immune subgroup:viral antigen IL-13 levels at 7 days, 14 days, 28 days and 3 months booster vaccination. (ELISpot assay)
Cellular immune subgroup:viral antigen IFN-γ levels | 7 days, 14 days, 28 days and 3 months after vaccination or placebo
  Cellular immune subgroup:viral antigen IFN-γ levels at 7 days, 14 days, 28 days and 3 months booster vaccination. (ELISpot assay)
Cross-neutralization subgroup:the cross-neutralizing ability of serum neutralizing antibodies in subjects. | 14 days, 28 days after vaccination or placebo
  The cross-neutralizing ability of serum neutralizing antibodies collected 14 days and 28 days after booster vaccination in the cross neutralization subgroup.
The immunological correlation of risk and protection against symptomatic COVID-19 and SARS-CoV-2 infection after booster vaccination. | after vaccination or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Fan Zhang, Study Director — AIM Vaccine Co., Ltd.
Locations (1):
- Sindh Infectious Diseases Hospital & Research Center Dow University of Health Sciences, Islamabad, Pakistan